CLINICAL TRIAL: NCT05877066
Title: Generating Real-world Ambispective Data to Study Participant Treatment Outcomes for Dupuytren's Contracture
Brief Title: Real-World Data Study to Understand Participant Treatment Outcomes for Dupuytren's Contracture
Acronym: GRASP-DC
Status: Terminated | Type: Observational
Why Stopped: Endo determined to discontinue its registries and the GRASP registry enrollment has been closed.
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Pulse Infoframe (Industry)
Responsible Party: Sponsor
Other Study IDs: EP01REG
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Dupuytren's Contracture
Keywords: Real world data; Retrospective; Prospective; Registry
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years

SUMMARY:
This is an observational study, meaning participants will not receive any investigational treatment as part of this study.

Researchers will collect real-world data (RWD), based on usual care, to gain a more in-depth knowledge of the natural history and the treatment outcomes of Dupuytren's Contracture (DC) to evaluate the management of DC.

DETAILED DESCRIPTION:
Each participant of the study will have their data collected from the date of confirmed diagnosis of DC to the date of enrollment in the registry, post consent. Data will be collected from the participants clinical records as well as from the participant directly. Data will be collected through Pulse Infoframe's technology platform.

ELIGIBILITY:
Key Inclusion Criteria:

* Any adult with a confirmed clinical diagnosis of DC.
* Age 18 years (or age of majority in their jurisdiction) or older at time of enrollment.
* Willing to participate in the registry (including completion of ePROs) and complete the informed consent form.
* Having received DC treatment, either non-surgical or surgical, within 2 weeks before enrollment, at enrollment or any time after the date of enrollment or not having received DC treatment after confirmed diagnosis of DC.
* Able to participate in English based registry.

Key Exclusion criteria:

* Not having a clinical diagnosis of DC.
* Age less than 18 years.
* Do not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of DC will be enrolled in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-02-26 (Actual)

PRIMARY OUTCOMES:
Number of Participants Receiving Each Treatment Type for DC | Up to 36 months

SECONDARY OUTCOMES:
Change from Baseline in Michigan Hand Questionnaire (MHQ) Scale Score | Up to 36 months
Change from Baseline in European Quality of Life Five Dimension (EQ-5D) Questionnaire Score | Up to 36 months
Change from Baseline in Unité Rhumatologique des Affections de la Main (URAM) Scale Score | Up to 36 months
Participant Satisfaction Questionnaire | Up to 36 months
Number of Participants Receiving Post-Procedural Care by the Treating Physician | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Information, Study Director — Endo Pharmaceuticals
Locations (7):
- United States (7):
  - Endo Pharmaceuticals Clinical Site 6, Phoenix, Arizona
  - Endo Pharmaceuticals Clinical Site 5, Greenwich, Connecticut
  - Endo Pharmaceuticals Clinical Site 4, Temple Terrace, Florida
  - Endo Pharmaceuticals Clinical Site 2, Indianapolis, Indiana
  - Endo Pharmaceuticals Clinical Site 1, Eatontown, New Jersey
  - Endo Pharmaceuticals Clinical Site 7, Charlotte, North Carolina
  - Endo Pharmaceuticals Clinical Site 3, Bend, Oregon